CLINICAL TRIAL: NCT02954107
Title: Longitudinal Early Epilepsy Study
Acronym: LEES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Epilepsiecentrum Kempenhaeghe (Industry)
Responsible Party: Sponsor
Other Study IDs: NL55455.068.15; 152055 (Other: Maastricht University Medical Centre+)
Record Dates: First submitted 2016-09-26; First posted 2016-11-03 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Absence Epilepsy; Epilepsy, Absence
MeSH Terms: conditions — Epilepsy, Absence | interventions — Videotape Recording; Neuropsychological Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Absence epilepsy: Children aged 6-12 years of age primarily presenting with episodes of brief loss of consciousness (absences) in an otherwise normal child in the previous 2 years. With an EEG showing 3 Hz (2.5-4.5 Hz) generalized rhythmic spike-and-wave complexes with a discharge duration of at least 3 seconds on a present or former EEG.
  Interventions: Other: MRI; Other: 24h-EEG + video; Other: Neuropsychological tests
- Controls: Overall healthy children aged 6-12 years of age following a regular school without major problems.
  Interventions: Other: MRI; Other: Neuropsychological tests

INTERVENTIONS:
Other: MRI
Other: 24h-EEG + video
  Groups: Absence epilepsy
Other: Neuropsychological tests

SUMMARY:
This longitudinal study will focus on the cognitive and brain development of children with absence epilepsy. In addition, the investigators aim to identify prognostic factors for cognitive deterioration and/or poor seizure control in these children.

DETAILED DESCRIPTION:
The aim is to study the cognitive and brain development of children with absence epilepsy. In addition, this study aims to identify prognostic factors for cognitive deterioration and/or poor seizure control.

Objective:

1. To study the development of cognition in children with absence epilepsy and the functional brain organization over time.
2. To find prognostic factors in terms of clinical, 24h-video-EEG or/and MRI characteristics for cognitive deterioration and/or poor seizure control in patients with absence epilepsy.

Study design:

2 year prospective longitudinal, controlled, comparative, clinical, follow up.

Study population:

60 children with recently diagnosed (<2 years) absence epilepsy, aged 6 to 12 years. In addition, this study includes a control group of 15 age and gender matched healthy volunteers.

Main study parameters/endpoints:

Endpoints are the development of clinical parameters (semiology, 24h-video-EEG and seizure control), neuropsychological/behavioural outcomes, structural/functional MRI parameters, and educational performance.

ELIGIBILITY:
Inclusion Criteria:

1. Primarily presented with daily occurring episodes of brief loss of consciousness (absences) in an otherwise normal child in the previous 2 years.
2. An EEG showing 3 Hz (2.5-4.5 Hz) generalized rhythmic spike-and-wave complexes with a discharge duration of at least 3 seconds on a present or former EEG(58).
3. Early absence epilepsy , defined as a confirmed diagnosis or seizures within 2 years.
4. Aged 6-12 years
5. Permitted accompanying factors:

   * A few generalized tonic-clonic seizures (assessed individually according to International League Against Epilepsy [ILAE] statements;
   * Mild myoclonic eye(lid) movements
   * Co-morbidities: Attention deficiency/concentration disorders, autism, dyslexia and anxiety. These do not form exclusion criteria as this is frequently seen in children with absence seizures and it might be uncertain if the co-morbidity is a manifestation of the absence epilepsy.

Exclusion Criteria:

* A potential subject (both for the control and patient group) who meets any of the following criteria will be excluded from participation in this study:

  * A diagnosis according to ILAE criteria of the following epilepsy syndromes: Juvenile Absence Epilepsy; Eyelid myoclonia with absences; Dravet syndrome; Epilepsy with myoclonic-atonic seizures; Epilepsy with Myoclonic Absences; Lennox-Gastaut syndrome; Frontal Lobe Epilepsy or other focal epilepsy.
  * A confirmed diagnosis of epilepsy/seizures for more than 2 years (59).
  * Recent hospitalizations in the last months or a history which might limit participation in or completion of the study protocol.
  * Behavioural characteristics which might hamper the gathering of useful MRI data.
  * Intellectual disability or other diseases/causes that may underlie cognitive impairment (i.e. neurodegenerative diseases).
  * History of major head trauma or head/brain surgery.
  * MRI lesions on (previous) structural brain MRI- or CT-scans or symptomatic epilepsies (e.g. epilepsy related to tumours, vascular abnormalities, congenital dysgenesia).
  * MRI contra-indications: claustrophobia, anxiety for an MRI scan, or presence of metallic objects (e.g. prostheses, pacemakers, metal clips on blood vessels, metal parts in the eye). Dental braces are no exclusion criterion for absence patients.
  * Regularly using drugs of abuse (asked during screening session).
  * Parents or participants (aged≥12 years) not willing to provide informed consent.
  * Parents or participants (aged≥12 years) who do not want to get informed whenever structural abnormalities are found during imaging.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 1. Children aged 6-12 years of age primarily presenting with episodes of brief loss of consciousness (absences) in an otherwise normal child in the previous 2 years. With an EEG showing 3 Hz (2.5-4.5 Hz) generalized rhythmic spike-and-wave complexes with a discharge duration of at least 3 seconds on a present or former EEG.
  2. Overall healthy children aged 6-12 years of age following a regular school without major problems.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Change of multimodal MRI parameters on brain connectivity | Baseline; first year; second year
Change of cognition measured by a battery of neuropsychological tests | Baseline; first year; second year
Time in months since start of medication till seizure control is attained, as assessed by anamnesis and a confirmatory routine-EEG. | Within 2 years

SECONDARY OUTCOMES:
Age in months at which seizures began (age of onset) assessed by interview at the baseline measurment | Baseline
Seizure semiology assessed by anamnesis and video-EEG | Baseline; first year; second year
  Seizure semiology will be re-assessed at the different time points
Epileptiform activity assessed by a 24h-EEG | Baseline; first year; second year
  Epileptiform acitivty will be re-assessed at the different time points

CONTACTS AND LOCATIONS:
Overall Officials: Johan SH Vles, MD, PHD, Study Director — Maastricht University Medical Center
Locations (2):
- Netherlands (2):
  - Kempenhaeghe, Heeze, Limburg
  - Maastricht University Medical Center, Maastricht, Limburg

IPD SHARING:
Plan to Share IPD: No